CLINICAL TRIAL: NCT05698849
Title: Effect of Amino Acid Addition to a Drink on the Appearance of Ingested Water in Body Fluids
Brief Title: Effect of Amino Acid Addition to a Drink on the Appearance of Ingested Water in Body Fluids (2859)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Entrinsic Beverage Company LLC (Unknown)
Responsible Party: Principal Investigator, Lewis James, Senior Lecturer in Nutrition, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LEON3151-2859
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2023-01

CONDITIONS: Rate of Water Appearance/Delivery in the Blood Water Balance

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, crossover design
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Commercially Available Sports Drink A (Placebo Comparator): A commercially available flavored electrolyte solution, The Coca-Cola Company
  Interventions: Other: Composition of Sports Drink
- Commercially Available Sports Drink B (Experimental): A commercially available flavored carbohydrate-electrolyte solution, PepsiCo
  Interventions: Other: Composition of Sports Drink
- Commercially Available Sports Drink A with added Amino Acids (Experimental): The same as sports drink A above (a commercially available flavored electrolyte solution, The Coca-Cola Company), but with the addition of a small amount of amino acids.
  Interventions: Other: Composition of Sports Drink

INTERVENTIONS:
Other: Composition of Sports Drink — The composition of sport drinks will be manipulated to determine the effect of drink composition on the appearance of ingested water in body fluid.

SUMMARY:
To determine the effects of a moderate amount of amino acids on the rate of water absorption and availability as a precursor fluid for sweat. Young and healthy (male or female) volunteers will take part in three experimental trials. In each trial, volunteers will be given one of two commercially available sports drinks or a commercially available sport drink with added amino acids in a double-blinded, randomised, crossover design. Each drink will be a single 550 mL bolus. All beverages will be labelled with deuterium (D2O). Trials will be compared for temporal accumulation of deuterium in plasma over the course of 60 minutes. Whole blood measurements of haemoglobin and haematocrit will also be made and plasma volume changes calculated. It is hypothesised that the amino acid trial will increase the rate of fluid absorption.

ELIGIBILITY:
Inclusion Criteria:

* Generally fit and healthy (determined by health screen questionnaire)
* Recreationally active (minimum 3 hours of physical activity per week including walking)

Exclusion Criteria:

* Any cardiovascular, gastrointestinal, renal or acute/chronic health conditions that may influence the outcomes
* Smoking (including vaping)
* BMI of greater than 30 (combined with a body fat percentage greater than 20%) or BMI lower than 17.5

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Time at which drink absorption rate was maximum (tmax) | 60 minutes
  Determined from D2O values in venous blood samples collected before and after drink ingestion
Maximum absorption of drink (Cmax) | 60 minutes
  Determined from D2O values in venous blood samples collected before and after drink ingestion
Area under the curve for D2O | 60 minutes
  Determined from D2O values in venous blood samples collected before and after drink ingestion

SECONDARY OUTCOMES:
Plasma volume | 60 minutes
  Determined from haemoglobin and haematocrit measures in venous blood samples collected before and after drink ingestion
Plasma osmolality | 60 minutes
  Determined from venous blood samples collected before and after drink ingestion
Urine specific gravity | 60 minutes
  Determined from urine samples collected before and after drink ingestion
Urine volume | Post-trial (at 60 minutes)
  Determined from urine samples collected after drink ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No